CLINICAL TRIAL: NCT03661801
Title: A Prospective Observational Study Examining the Clinical Utility of Novel Pleural Fluid, Biopsy and Serum Bio Markers for the Investigation of Pleural Effusions
Brief Title: Novel Pleural Fluid, Biopsy and Serum Biomarkers for the Investigation of Pleural Effusions
Acronym: INVEST
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Rocket Medical plc (Other)
Responsible Party: Sponsor
Other Study IDs: INVEST Version 1.0
Record Dates: First submitted 2018-09-04; First posted 2018-09-07 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Respiratory Disease; Pleural Effusion; Lung Cancer
Keywords: Respiratory; Pleural Effusion
MeSH Terms: conditions — Respiration Disorders; Pleural Effusion; Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For patients with undiagnosed pleural effusion or thickening, an extra 10ml blood and 10 ml fluid will be taken for study purposes when these samples are collected for clinical purposes. For these patients undergoing pleural biopsy, as part of their clinical care, an extra sample will be taken for the trial. For patients with suspected lung cancer, one extra biopsy sample will be taken when the participants have their diagnostic bronchoscopic biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to prospectively asses established biomarkers in the diagnosis and prognosis of patients and will include assessment of a number of biomarkers, genomics and proteomics.

DETAILED DESCRIPTION:
A prospective observation study examining the clinical utility of novel pleural fluid, biopsy and serum biomarkers for the investigation of pleural effusions (INVEST). The INVEST study will collect blood, pleural fluid and tissue samples from donors, allowing the opportunity to apply several novel blood and pleural fluid tests with interpretation of results in the context of clinical data and diagnostic suspicion. Through the prospective application of multiple tests, we aim to validate the sensitivity and specificity of existing biomarkers and identify novel markers that aid in the diagnostic pathway of pleural diseases. Because samples and data will be stored for future use, many other different tests, methods and techniques may be used in the future to provide information that we cannot foresee.

ELIGIBILITY:
Inclusion Criteria:

* Undiagnosed pleural effusion or pleural thickening requiring investigation by one of the following:

  * Pleural aspiration
  * Pleural biopsies from medical thoracoscopy or
  * Ultrasound guided biopsies as part of the clinical plan
* Suspected lung cancer undergoing bronchoscopy and biopsies.

Exclusion Criteria:

* Inability to give written informed consent
* Inability to obtain pleural fluid, blood, endobronchial or pleural biopsies as applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective single centre study looking to recruit 300 participants to help prospectively evaluate the sensitivity and specificity of known diagnostic biomarkers and discover novel biomarkers in pleural diseases. Patients aged 18 or over, requiring investigation and/or management of any undiagnosed pleural effusion or pleural thickening will be approached about the study within Oxford University Hospital NHS Foundation Trust.
Sampling Method: Non-Probability Sample
Enrollment: 313 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Protein expression levels of specific biomarkers | At enrolment
  All study samples will be analysed with specific laboratory based techniques (enzyme-linked immunosorbent assay, ELISA, or luminex assay.
  - Existing biomarkers will be prospectively evaluated based on the underlying disease:
  * Mesothelin
  * Procalcitonin
  * Brain natriuretic peptide
  * Fibulin
  * Osteopontin
  * ADA
  * additional markers will be included on the panel depending on the patient's underlying disease this could include inflammatory markers, cancer related peptides and immune cell profiling.
  The above tests have been demonstrated in the BTS Guidelines in pleural disease entitled "Investigation of a unilateral pleural effusion in adults" to have utility in the diagnosis of infectious, malignant, tuberculous and heart failure related effusion.
  Samples will also be processed for the identification of novel markers with diagnostic or therapeutic importance. Specific cell population will be measured with flow cytometry to detect the immune response of different

SECONDARY OUTCOMES:
The analysis of protein and gene expression profile in cell subpopulation of pleural fluid, pleural and endobronchial biopsies and blood samples. | At enrolment
  To correlate gene expression, immune sub population, protein levels with pleural disease prognoses

CONTACTS AND LOCATIONS:
Overall Officials: Najib Rahman, Principal Investigator — University of Oxford
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided